CLINICAL TRIAL: NCT05288894
Title: Multicenter Italian Registry From the Italian Pediatric Cardiology Society (SICP) Working Group (WG) on CMR/CT for the Repaired Tetralogy of Fallot
Brief Title: Repaired Tetralogy of Fallot Italian Registry
Acronym: RETE-Fallot
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Collaborators: SICP WG CMR/CT (Unknown); Fondazione Toscana Gabriele Monasterio (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Medical Doctor, Azienda Ospedaliero, Universitaria Ospedali Riuniti
Other Study IDs: SICP WG CMR/CT 001
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Tetralogy of Fallot; Cardiac Death, Sudden; Cardiac Arrhythmia; Cardiac Event
MeSH Terms: conditions — Tetralogy of Fallot; Death, Sudden, Cardiac; Arrhythmias, Cardiac; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Repaired Tetralogy of Fallot: A patient affected by Tetralogy of Fallot (right ventricle outflow obstruction, right ventricle hypertrophy, ventricular septal defect, aortic overriding of the ventricular defect) that already underwent cardiac surgery for the correction.
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance imaging — A routine cardiac magnetic resonance imaging with biventricular function evaluation, atrial volumes, LGE acquisitions, and pulmonary and aortic assesment.

SUMMARY:
The CMR/CT WG of the Italian pediatric cardiology society set up a multi-center observational clinical database of repaired-TOF evaluated. This registry will enroll prospectively patients evaluated by CMR for clinical indication in most of the CHD Italian centers. Data collection will include surgical history, clinical data, imaging data, and also adverse cardiac events for a period of 6 years.

DETAILED DESCRIPTION:
This is an observational prospective registry that will enroll patients presenting with repaired Tetralogy of Fallot (TOF) undergoing a cardiac magnetic resonance (CMR) imaging study in our recruiting CMR-Laboratories.

CMR imaging studies will include the evaluation of biventricular volumes and function, atrial volumes and function, and the Late Gadolinium Enhancement (LGE), along with the evaluation of the anatomy and flow of the main pulmonary arteries and branches. We will also assess the aortic valve for regurgitation and measurement of the aortic size.

At follow-up, any interventional or surgical procedures performed and symptoms or any major (Death) and cardiac (cardiac-related hospitalization) events will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Repaired - TOF

Exclusion Criteria:

* Age < 10 years
* Other associated complex pathology such as MAPCAs, Atrioventricular canal, Ebstein
* Incomplete CMR exam

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a repaired-TOF without associated complex pathology underwent CMR imaging.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac death | 6 years
  Number of Participants with cardiac-releted death

SECONDARY OUTCOMES:
Hospitalizations | 6 years
  Rate of cardiac-related hospitalizations due to cardiac arrhythmias or cardaio failure

CONTACTS AND LOCATIONS:
Locations (1):
- CCPC, Ancona, The Marches, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffman JI. Incidence of congenital heart disease: I. Postnatal incidence. Pediatr Cardiol. 1995 May-Jun;16(3):103-13. doi: 10.1007/BF00801907. PMID 7617503
- [Background] Villafane J, Feinstein JA, Jenkins KJ, Vincent RN, Walsh EP, Dubin AM, Geva T, Towbin JA, Cohen MS, Fraser C, Dearani J, Rosenthal D, Kaufman B, Graham TP Jr; Adult Congenital and Pediatric Cardiology Section, American College of Cardiology. Hot topics in tetralogy of Fallot. J Am Coll Cardiol. 2013 Dec 10;62(23):2155-66. doi: 10.1016/j.jacc.2013.07.100. Epub 2013 Sep 27. PMID 24076489
- [Background] Geva T. Repaired tetralogy of Fallot: the roles of cardiovascular magnetic resonance in evaluating pathophysiology and for pulmonary valve replacement decision support. J Cardiovasc Magn Reson. 2011 Jan 20;13(1):9. doi: 10.1186/1532-429X-13-9. PMID 21251297
- [Background] Geva T. Indications for pulmonary valve replacement in repaired tetralogy of fallot: the quest continues. Circulation. 2013 Oct 22;128(17):1855-7. doi: 10.1161/CIRCULATIONAHA.113.005878. Epub 2013 Sep 24. No abstract available. PMID 24065609
- [Background] Geva T, Sandweiss BM, Gauvreau K, Lock JE, Powell AJ. Factors associated with impaired clinical status in long-term survivors of tetralogy of Fallot repair evaluated by magnetic resonance imaging. J Am Coll Cardiol. 2004 Mar 17;43(6):1068-74. doi: 10.1016/j.jacc.2003.10.045. PMID 15028368
- [Background] Samad MD, Wehner GJ, Arbabshirani MR, Jing L, Powell AJ, Geva T, Haggerty CM, Fornwalt BK. Predicting deterioration of ventricular function in patients with repaired tetralogy of Fallot using machine learning. Eur Heart J Cardiovasc Imaging. 2018 Jul 1;19(7):730-738. doi: 10.1093/ehjci/jey003. PMID 29538684
- [Background] Wald RM, Valente AM, Gauvreau K, Babu-Narayan SV, Assenza GE, Schreier J, Gatzoulis MA, Kilner PJ, Koyak Z, Mulder B, Powell AJ, Geva T. Cardiac magnetic resonance markers of progressive RV dilation and dysfunction after tetralogy of Fallot repair. Heart. 2015 Nov;101(21):1724-30. doi: 10.1136/heartjnl-2015-308014. Epub 2015 Aug 14. PMID 26276804
- [Background] Gliklich RE, Dreyer NA, Leavy MB, editors. Registries for Evaluating Patient Outcomes: A User's Guide [Internet]. 3rd edition. Rockville (MD): Agency for Healthcare Research and Quality (US); 2014 Apr. Report No.: 13(14)-EHC111. Available from http://www.ncbi.nlm.nih.gov/books/NBK208616/ PMID 24945055
- [Background] Trojano M. Can databasing optimise patient care? J Neurol. 2004 Sep;251 Suppl 5:v79-v82. doi: 10.1007/s00415-004-1513-x. PMID 15549361
- [Background] Ravaglioli A, Ait-Ali L, Federici D, Salvadori S, Pllumi A, Pak V, Marrone C, Pizzuto A, Bonhoeffer P, Festa P. The impact of native Fallot anatomy on future therapeutic requirements and outcomes at follow-up. Cardiovasc Ultrasound. 2021 Jun 19;19(1):23. doi: 10.1186/s12947-021-00249-y. PMID 34147117
- [Background] Clemente EA, Casares AP, Frontera PR, Calvar JMC, de Toledo JS. Finding the Optimal Timing for Repair of Standard Tetralogy of Fallot: Analysis of Cardiac Magnetic Resonance and Echocardiography Parameters Related to Intermediate Term Outcomes in a Pediatric Population. Pediatr Cardiol. 2021 Aug;42(6):1324-1333. doi: 10.1007/s00246-021-02615-z. Epub 2021 May 2. PMID 33934202
- [Background] Egbe AC, Kothapalli S, Borlaug BA, Ammash NM, Najam M, Bajwa N, Tarek K, Mathew J, Connolly HM. Mechanism and Risk Factors for Death in Adults With Tetralogy of Fallot. Am J Cardiol. 2019 Sep 1;124(5):803-807. doi: 10.1016/j.amjcard.2019.05.048. Epub 2019 Jun 7. PMID 31272701
- [Background] Bokma JP, Winter MM, Vehmeijer JT, Vliegen HW, van Dijk AP, van Melle JP, Meijboom FJ, Post MC, Zwinderman AH, Mulder BJ, Bouma BJ. QRS fragmentation is superior to QRS duration in predicting mortality in adults with tetralogy of Fallot. Heart. 2017 May;103(9):666-671. doi: 10.1136/heartjnl-2016-310068. Epub 2016 Nov 1. PMID 27803032
- [Background] Berul CI, Hill SL, Geggel RL, Hijazi ZM, Marx GR, Rhodes J, Walsh KA, Fulton DR. Electrocardiographic markers of late sudden death risk in postoperative tetralogy of Fallot children. J Cardiovasc Electrophysiol. 1997 Dec;8(12):1349-56. doi: 10.1111/j.1540-8167.1997.tb01031.x. PMID 9436772
- [Background] Valente AM, Cook S, Festa P, Ko HH, Krishnamurthy R, Taylor AM, Warnes CA, Kreutzer J, Geva T. Multimodality imaging guidelines for patients with repaired tetralogy of fallot: a report from the AmericanSsociety of Echocardiography: developed in collaboration with the Society for Cardiovascular Magnetic Resonance and the Society for Pediatric Radiology. J Am Soc Echocardiogr. 2014 Feb;27(2):111-41. doi: 10.1016/j.echo.2013.11.009. No abstract available. PMID 24468055
- [Background] Toyono M, Harada K, Tamura M, Yamamoto F, Takada G. Myocardial acceleration during isovolumic contraction as a new index of right ventricular contractile function and its relation to pulmonary regurgitation in patients after repair of tetralogy of Fallot. J Am Soc Echocardiogr. 2004 Apr;17(4):332-7. doi: 10.1016/j.echo.2003.12.022. PMID 15044866
- [Background] Stout KK, Daniels CJ, Aboulhosn JA, Bozkurt B, Broberg CS, Colman JM, Crumb SR, Dearani JA, Fuller S, Gurvitz M, Khairy P, Landzberg MJ, Saidi A, Valente AM, Van Hare GF. 2018 AHA/ACC Guideline for the Management of Adults With Congenital Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Apr 2;73(12):e81-e192. doi: 10.1016/j.jacc.2018.08.1029. Epub 2018 Aug 16. No abstract available. PMID 30121239
- [Background] Diller GP, Dimopoulos K, Okonko D, Li W, Babu-Narayan SV, Broberg CS, Johansson B, Bouzas B, Mullen MJ, Poole-Wilson PA, Francis DP, Gatzoulis MA. Exercise intolerance in adult congenital heart disease: comparative severity, correlates, and prognostic implication. Circulation. 2005 Aug 9;112(6):828-35. doi: 10.1161/CIRCULATIONAHA.104.529800. Epub 2005 Aug 1. PMID 16061735
- [Background] Baumgartner H, De Backer J, Babu-Narayan SV, Budts W, Chessa M, Diller GP, Lung B, Kluin J, Lang IM, Meijboom F, Moons P, Mulder BJM, Oechslin E, Roos-Hesselink JW, Schwerzmann M, Sondergaard L, Zeppenfeld K; ESC Scientific Document Group. 2020 ESC Guidelines for the management of adult congenital heart disease. Eur Heart J. 2021 Feb 11;42(6):563-645. doi: 10.1093/eurheartj/ehaa554. No abstract available. PMID 32860028
- [Background] Festa P, Ait-Ali L, Prontera C, De Marchi D, Fontana M, Emdin M, Passino C. Amino-terminal fragment of pro-brain natriuretic hormone identifies functional impairment and right ventricular overload in operated tetralogy of Fallot patients. Pediatr Cardiol. 2007 Sep-Oct;28(5):339-45. doi: 10.1007/s00246-007-0009-8. Epub 2007 Jun 29. PMID 17607499
- [Background] Heng EL, Bolger AP, Kempny A, Davlouros PA, Davidson S, Swan L, Uebing A, Pennell DJ, Gatzoulis MA, Babu-Narayan SV. Neurohormonal activation and its relation to outcomes late after repair of tetralogy of Fallot. Heart. 2015 Mar;101(6):447-54. doi: 10.1136/heartjnl-2014-306398. Epub 2014 Oct 28. PMID 25351509